CLINICAL TRIAL: NCT03123432
Title: Combination of Arginine, Glutamine, and Omega-3 Fatty Acid Supplements for Perioperative Enteral Nutrition in Surgical Patients With Gastric Adenocarcinoma or Gastrointestinal Stromal Tumor (GIST)
Brief Title: Immunomodulating Nutrients in Perioperative Patients With Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jaw-Yuan Wang, MD, PhD, Professor, Vice Superintendent, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-2011-05-01(II)
Record Dates: First submitted 2017-04-05; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Gastric Cancer
Keywords: immunomodulating nutrients
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- immunomodulating nutrients enriched diet (Experimental): Patients received oral feeding with an ordinary diet plus 400 mL/day (400 kcal/day) of the immunomodulating nutrients enriched diet for 3-5 days before curative surgery for gastric adenocarcinoma or gastric GIST. On postoperative day 3, enteral nutrition (EN) was initiated with 5% glucose in water at a rate of 20 mL/h. On postoperative day 4, patients received a semi-liquid diet plus 400 mL/day (400 kcal/day) of the immunomodulating nutrients enriched diet. From postoperative day 5-14 or to discharge whichever occurred first, 1200 mL/day (1200 kcal/day) of the interventional diet was administered, and an oral soft diet was also administered if no postoperative complications developed and if oral feeding was not prohibited.
  Interventions: Dietary Supplement: immunomodulating nutrients enriched diet
- standard diet (Active Comparator): Patients received oral feeding with an ordinary diet plus 400 mL/day (400 kcal/day) of the standard diet for 3-5 days before curative surgery for gastric adenocarcinoma or gastric GIST. On postoperative day 3, EN was initiated with 5% glucose in water at a rate of 20 mL/h. On postoperative day 4, patients received a semi-liquid diet plus 400 mL/day (400 kcal/day) of the interventional diet. From postoperative day 5-14 or to discharge whichever occurred first, 1200 mL/day (1200 kcal/day) of the standard diet was administered, and an oral soft diet was also administered if no postoperative complications developed and if oral feeding was not prohibited.
  Interventions: Dietary Supplement: standard diet

INTERVENTIONS:
Dietary Supplement: immunomodulating nutrients enriched diet
  Other Names: neo-mune
  Arms: immunomodulating nutrients enriched diet
Dietary Supplement: standard diet
  Arms: standard diet

SUMMARY:
The survey is a phase IV, prospective randomized clinical trial to determine whether an immunomodulating nutrient-enriched diet compared to a standard diet can improve nutritional status and reduce postoperative infection and surgery-induced immune suppression in patients with gastric cancer or GIST undergoing major surgery in a single medical center.

DETAILED DESCRIPTION:
Primary Objective:

1. The primary end points:

   To evaluate the effect of immunomodulating diets on the postoperative inflammatory response: including interleukin (IL)-6, C-reactive protein (CRP), and tumor necrosis factor-α (TNF-α).
2. Secondary Objectives:

(1). Biochemistry parameters: glucose,blood urine nitrogen, creatinine, aspartate aminotransferase, alanine aminotransferase, triglycerides, cholesterol, low-density lipoprotein, high-density lipoprotein, sodium, and leukocyte count.

(2). Nutritional status: albumin, prealbumin, BMI (3). Adverse events (4). Clinical outcomes: postoperative complications, time to first bowel action and length of hospital stay after surgery.

Number of Subjects: Eligible patients will be randomized in 2 arms in the ratio of 1:1, to reach 15 patients at least in each.

Plan of the Study:

1. This is a randomized, comparative, double blinded study in 2 arms.
2. Study Schedule Study date: the time getting approval letter issued by both regulatory authority and institutional review board (IRB). Duration of the study: 5 years.
3. Duration of Treatment: Treatment was administered before curative surgery for gastric adenocarcinoma or gastric GIST, and postoperative day 5-14 or to discharge whichever occurred first, or consent withdrawal during any time of the study, when the patient would be withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-85 years old
* Histologically proven primary gastric cancer or GIST.
* Patients was planning to receive elective curative gastric surgery, such as partial gastrectomy, subtotal gastrectomy, proximal gastrectomy, total gastrectomy, etc.
* Patient is able to understand the requirements of the study and written informed consent was obtained from each subject.

Exclusion Criteria:

* They were less than 20 years or over 85 years old
* Hepatic dysfunction or bile stasis (serum total bilirubin >2.5 mg/dL)
* Renal dysfunction (serum creatinine >1.5 mg/dL), or required hemodialysis
* Cardiac dysfunction (NYHA functional class >III, or stroke history)
* Severe hypoalbuminemia (albumin <2.5 g/dL)
* Karnofsky performance status less than 60
* Overweight (body mass index [BMI] >30 kg/m2)
* Exhibited drug abuse or chronic alcoholism
* Had life-threatening disease, or underwent emergent surgery
* With infection or bowel obstruction
* Pregnant or lactating
* Had received chemotherapy within 14 days of the initiation of the trial
* Had received immunosuppressive therapy or had immunological diseases recently
* Had already participated in another clinical study with an investigational drug or an investigational medical device within a month of the initiation or during the study
* Hypersensitive to casein, fish oil, soybean, or corn oil

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
immunomodulating effects | at discharge from the hospital or 14 days after surgery, whichever occurred first
  Inflammatory markers including interleukin (IL)-6, C-reactive protein (CRP), and tumor necrosis factor-α (TNF-α) were employed to assess inflammatory processes.

SECONDARY OUTCOMES:
blood glucose | at discharge from the hospital or 14 days after surgery, whichever occurred first
blood urine nitrogen | at discharge from the hospital or 14 days after surgery, whichever occurred first
blood aspartate aminotransferase (AST) in U/L | at discharge from the hospital or 14 days after surgery, whichever occurred first
blood alanine aminotransferase (ALT) in U/L | at discharge from the hospital or 14 days after surgery, whichever occurred first
blood triglycerides (TG) in mg/dL | at discharge from the hospital or 14 days after surgery, whichever occurred first
blood cholesterol in mg/mL | at discharge from the hospital or 14 days after surgery, whichever occurred first
blood low-density lipoprotein (LDL) in mg/mL | at discharge from the hospital or 14 days after surgery, whichever occurred first
blood high-density lipoprotein (HDL) in mg/mL | at discharge from the hospital or 14 days after surgery, whichever occurred first
blood sodium (Na) mEq/L | at discharge from the hospital or 14 days after surgery, whichever occurred first
blood leukocyte count cells/μL | at discharge from the hospital or 14 days after surgery, whichever occurred first
blood albumin in g/dL | at discharge from the hospital or 14 days after surgery, whichever occurred first
blood prealbumin in mg/dL | at discharge from the hospital or 14 days after surgery, whichever occurred first
body mass index (BMI) in kg/m^2 | at discharge from the hospital or 14 days after surgery, whichever occurred first
postoperative complications | at discharge from the hospital or 14 days after surgery, whichever occurred first
  postoperative complications that related to surgery
time to first bowel action | at discharge from the hospital or 14 days after surgery, whichever occurred first
  interval of surgery to first bowel action (hours)
length of hospital stay after surgery | at discharge from the hospital or 14 days after surgery, whichever occurred first
  length of hospital stay after surgery (days)

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Yuan Wang, PhD, Study Chair — Division of Colorectal Surgery, Department of Surgery, Kaohsiung Medical University Hospital, Kaohsiung Medical University
Locations (1):
- Chung-Ho Memorial Hospital, Kaohsiung Medical University:, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No